CLINICAL TRIAL: NCT05806398
Title: Use of a Glass Ionomer Sealant in First Permanent Molars Affected by Molar Incisor Hypomineralization
Brief Title: Use of a Glass Ionomer Sealant in Molar Incisor Hypomineralization
Status: Recruiting | Type: Observational
Sponsor: IRCCS Burlo Garofolo (Other)
Responsible Party: Sponsor
Other Study IDs: RC 50/22
Record Dates: First submitted 2023-03-28; First posted 2023-04-10 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Molar Incisor Hypomineralization
Keywords: Molar Incisor Hypomineralization (MIH) Molars; Glass ionomer sealant; Prevention
MeSH Terms: conditions — Molar Hypomineralization

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Molar Incisor Hypomineralization (MIH) is a worldwide widespread qualitative developmental defect of the dental enamel with a multifactorial aetiology defined in 2001 as an "hypomineralization of systemic origin affecting one or more permanent molars, usually first permanent molars (FPMs), with or without the involvement of one or more affected permanent incisors". Clinically MIH lesions appear as demarcated opacities with a creamy-white to yellow-brown colour depending on the severity of the defect that is classified as mild or severe (levels of severity) according to the European Academy of Pediatric Dentistry (EAPD) severity criteria. The distribution of the lesions is asymmetrical and their severity varies from a patient to another and also within the mouth of the same patient. Due to its porous structure with an altered prism organization and an increased content of proteins, the hypomineralized enamel has reduced mechanical properties and a lower refractive index if compared to the sound enamel. MIH is associated to a large number of objective and subjective problems as an altered aesthetics, an increased risk of plaque accumulation, caries, post-eruptive breakdown (PEB), reduced retention rates of adhesive materials, hypersensitivity and difficulty in anesthetizing the affected teeth making its management a challenging condition. Among preventive measures, pit-and-fissure sealants are a valuable and effective treatment to prevent occlusal caries in FPMs when they are still intact. However, since their efficacy is closely related to the sealant retention, they have to be monitored over time. When the molar to be sealed is fully erupted and isolation is adequate, resin-based sealants are indicated while if the moisture control is inadequate and/or the tooth is hypersensitive and patient is not sufficiently cooperative, low-viscous glass ionomer cements (GICs) are suggested as a temporary measure until the eruption is completed and both symptoms and cooperation are improved. To date, the scientific knowledge regarding the use of different type of sealants in MIH affected molars is insufficient to draw exhaustive conclusions and further studies are needed to deepen the knowledge on this topic. The aim of this study is to assess, by clinical examination, the survival rate of a glass ionomer sealant in MIH affected FPMs at 12 months of follow-up.

DETAILED DESCRIPTION:
Molar Incisor Hypomineralization (MIH) is a worldwide widespread qualitative developmental defect of the dental enamel with a multifactorial aetiology defined in 2001 as an "hypomineralization of systemic origin affecting one or more permanent molars, usually first permanent molars (FPMs), with or without the involvement of one or more affected permanent incisors". Clinically MIH lesions appear as demarcated opacities with a creamy-white to yellow-brown colour depending on the severity of the defect that is classified as mild or severe (levels of severity) according to the European Academy of Pediatric Dentistry (EAPD) severity criteria. The distribution of the lesions is asymmetrical and their severity varies from a patient to another and also within the mouth of the same patient. Due to its porous structure with an altered prism organization and an increased content of proteins, the hypomineralized enamel has reduced mechanical properties and a lower refractive index if compared to the sound enamel. MIH is associated to a large number of objective and subjective problems as an altered aesthetics, an increased risk of plaque accumulation, caries, post-eruptive breakdown (PEB), reduced retention rates of adhesive materials, hypersensitivity and difficulty in anesthetizing the affected teeth making its management a challenging condition.

Considering MIH histopathological features, while for incisors lesions are mainly an aesthetic issue, for molars they represent a real functional problem. Being FPMs subjected to higher masticatory loads than incisors and being located backward in the mouth, they have an increased risk of plaque accumulation, caries, PEB and are more difficult to be properly brushed especially if hypersensitive. An early diagnosis based on the EAPD judgement criteria and prevention are fundamental for acting with a minimally invasive therapeutic approach gaining the patient's cooperation and avoiding the most frequent related issues. Among preventive measures, pit-and-fissure sealants are a valuable and effective treatment to prevent occlusal caries in FPMs when they are still intact. However, since their efficacy is closely related to the sealant retention, they have to be monitored over time. When the molar to be sealed is fully erupted and isolation is adequate, resin-based sealants are indicated while if the moisture control is inadequate and/or the tooth is hypersensitive and patient is not sufficiently cooperative, low-viscous glass ionomer cements (GICs) are suggested as a temporary measure until the eruption is completed and both symptoms and cooperation are improved. About the use of resinous sealants in MIH molars, to date, literature data are limited and debated. About the use of glass ionomer (GI) sealants, several studies have been performed on sound molars but only a few on MIH molars. If the GI sealants' self-adhesive features, their high fluoride-release, hydrophilic properties and simple use are well known, their bond strength to the hypomineralized enamel and the survival rates on MIH molars are still controversial. To date, the scientific knowledge regarding the use of different type of sealants in MIH affected molars is insufficient to draw exhaustive conclusions and further studies are needed to deepen the knowledge on this topic. The aim of this study is to assess, by clinical examination, the survival rate of a glass ionomer sealant in MIH affected FPMs at 12 months of follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. FPMs of children aged between 6 and 10 years;
2. Erupted MIH affected FPMs presenting lesions on the occlusal surface;
3. Good general health conditions;
4. Sufficient cooperative behaviour;
5. Signature of the informed consent to the study by patients' parents or by their legal guardians

Exclusion Criteria:

1. FPMs presenting fluorosis, amelogenesis imperfecta, white spots, or other enamel defects that are in differential diagnosis with MIH;
2. FPMs presenting the occlusal surface already sealed or restored;
3. FPMs presenting occlusal cavitated caries (ICDAS Pit and Fissures ≥ 3)
4. FPMs presenting severe PEB involving the dentin;
5. Children with orthodontic devices hiding FPMs.

Ages: 6 Years to 10 Years | Sex: All
Age Groups: Child
Study Population: Children aged between 6 and 10 years with erupted MIH affected FPMs presenting lesions on the occlusal surface
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Glass ionomer sealant survival rate | At 12-month follow up
  Percentage of satisfactory status sealant in FPMs affected by MIH

CONTACTS AND LOCATIONS:
Overall Officials: Milena Cadenaro, MD, Study Director — IRCCS materno infantile Burlo Garofolo
Locations (1):
- IRCCS Burlo Garofolo, Trieste, Italy